CLINICAL TRIAL: NCT05900765
Title: A Multicenter, Open-label Phase II Study on the Treatment of Newly Diagnosed Early-stage Hodgkin's Lymphoma With Zimberelimab (GLS-010) Combined With AVD Regimen (Doxorubicin, Vindesine, Dacarbazine) Under the Guidance of PET/CT
Brief Title: A Study of Zimberelimab(GLS-010) Combined With AVD for Newly Diagnosed Early-stage Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Li Zhiming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-134-01
Record Dates: First submitted 2023-06-02; First posted 2023-06-13 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Zimberelimab; PD-1 Checkpoint Inhibitor; AVD
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zimberelimab combined with or without AVD sequential radiotherapy (Experimental): 1. Combination therapy： Subjects received Zimberelimab 240mg Q3W 2 cycle.
     According to the results of PET/CT evaluation:
     CR: Additional 2 cycles of Zimberelimab (4 cycles of Zimberelimab monotherapy in total); PR: 2 cycles of Zimberelimab+ AVD therapy (only PR patients combined with AVD). Subjects who did not achieve a Partial Response (PR) or Complete Response (CR) in their initial or subsequent efficacy evaluations, and whose potential for benefit was deemed unlikely by the investigator, were discontinued from the study.
  2. Radiotherapy treatment period (patients with CR/PR): Sequentially radiation therapy 20-30Gy.
  Interventions: Drug: Zimberelimab 240mg

INTERVENTIONS:
Drug: Zimberelimab 240mg — AVD regimen:
  Doxorubicin 25mg/m2, d1, d15, IV; Vincristine 3mg/m2, d1, d15 IV; Dacarbazine 0.375mg/m2, d1, d15 IV
  Other Names: GLS-010

SUMMARY:
This is a multicenter, open-label single-arm phase II study to evaluate the efficacy and safety of Zimberelimab (GLS-010) combined with AVD for newly diagnosed early-stage Hodgkin's lymphoma under the guidance of PET/CT.

DETAILED DESCRIPTION:
Despite achieving good disease control and long-term survival rates for over 80% of classical Hodgkin lymphoma (cHL) patients who receive first-line therapy, approximately 10% of early-stage and 30% of advanced cHL patients experience disease relapse or refractoriness after initial treatment, and only half of the patients can be cured through high-dose therapy (HDT) and autologous stem cell transplantation (ASCT). Meanwhile, the current standard first-line treatment still centers around conventional chemotherapy with cytotoxic agents. As such, the clinical challenge of cHL first-line treatment lies in striking a balance between efficacy and toxicity, and developing low-toxicity, high-efficiency treatment strategies to achieve the optimal treatment goal of maximizing efficacy while minimizing short- and long-term toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with primary classical Hodgkin lymphoma (HL) based on histopathology.
2. Stage I-II .
3. At least one measurable target lesion（Lugano 2014）.
4. Age 18 years or older (including 18 years) to 45 years (recent fertility requirements and concern about chemotherapy side effects), or age >60 years (older patients who are frail and unwilling to undergo chemotherapy), male or female.
5. ECOG PS 0-3,
6. Expected survival ≥ 3 months.

Exclusion Criteria:

1. Hodgkin's lymphoma with nodular lymphocyte predominant type.
2. Patients who are scheduled to undergo subsequent autologous stem cell transplantation.
3. Contraindications to radiotherapy.
4. With central nervous system (meningeal or parenchymal) involvement.
5. Contraindications to immune checkpoint inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) after 2 cycles | Up to approximately 2 months
  Percentage of the sum of the number of patients in complete remission (CR), complete remission without confirmation (CRu) to the total number of patients in the full analysis set

SECONDARY OUTCOMES:
Objective response rate (ORR) after 4 cycles ( Lugano2014) | Up to approximately 2 years
  ORR is proportion of subjects with complete response(CR) or partial response(PR)
Complete response rate (CRR) after 4 cycles ( Lugano2014) | Up to approximately 2 years
  Percentage of the sum of the number of patients in complete remission (CR), complete remission without confirmation (CRu) to the total number of patients in the full analysis set
Total ORR and CRR after Zimberelimab treatment + radiotherapy | Up to approximately 2 years
  ORR is proportion of subjects with complete response(CR) or partial response(PR); Percentage of the sum of the number of patients in complete remission (CR), complete remission without confirmation (CRu) to the total number of patients in the full analysis set
Duration of response (DOR) | Up to approximately 2 years
  Duration of response (DoR) is defined as the period from the first documentation of confirmed response (CR or PR) to the first documentation of progressive disease(PD) or death due to any cause, whichever occurs first
Progression-free survival time (PFS) | Up to approximately 2 years
  Progression-free survival (PFS) is defined as the time from the first dose of investigational products until documentation of PD or death due to any cause, whichever occurs first
Overall survival (OS) | Up to approximately 2 years
  Overall survival (OS) is defined as the time from the first dose of investigational products until death due to any cause
Incidence and severity of adverse events(AEs) | Up to approximately 2 years
  Incidence and severity of AEs is aim to evaluate the safety of Zimberelimab(GLS-010) Combined With AVD

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No